CLINICAL TRIAL: NCT02467907
Title: A Multicenter Open-Label Single-Arm Phase II Study Evaluating the Safety and Efficacy of Bevacizumab in Combination With Carboplatin and Paclitaxel in Patients With Metastatic, Recurrent or Persistent Cervical Cancer
Brief Title: Safety and Efficacy of Bevacizumab in Combination With Carboplatin and Paclitaxel for Metastatic, Recurrent or Persistent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO29594; 2014-005491-28 (EudraCT Number)
Record Dates: First submitted 2015-05-21; First posted 2015-06-10 (Estimated); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Bevacizumab; Carboplatin; Paclitaxel

ARMS (1):
- Bevacizumab in Combination with Carboplatin and Paclitaxel (Experimental): Administration of bevacizumab, carboplatin and paclitaxel once every 3 weeks, for at least 6 cycles, until disease progression (as assessed by the investigator), unacceptable toxicity, physician or participant decision or withdrawal of consent. If either chemotherapy or bevacizumab is discontinued, the participant may continue to receive the other ongoing therapy.
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — Intravenous (i.v.) administration of 15 mg/kg bevacizumab once every 3 weeks
  Other Names: Avastin, RO4876646
Drug: Carboplatin — Administration of carboplatin at 5 milligrams per milliliter*minute (mg/mL*min) on Day 1 every 3 weeks for at least 6 cycles
Drug: Paclitaxel — Administration of paclitaxel at a dose of 175 milligrams per square meter (mg/m^2) on Day 1 every 3 weeks for at least 6 cycles

SUMMARY:
This study is to assess safety as defined by the frequency and severity of gastrointestinal (GI) perforation/fistula, GI-vaginal fistula and genitourinary (GU) fistula in participants treated with bevacizumab 15 milligrams per kilogram (mg/kg) in combination with paclitaxel and carboplatin, all repeated every 3 weeks, for recurrent, persistent or metastatic cervical cancer. In addition, this study will include evaluation of the overall safety profile of bevacizumab in combination with paclitaxel and carboplatin in this setting, assessment of GI perforation/fistula, GI-vaginal fistula and GU fistula events over time, and evaluation of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Life expectancy greater than or equal to (>=3) months
* For women who are not postmenopausal or surgically sterile, agreement to remain abstinent or use single or combined contraceptive methods that result in a failure rate of less than (<) 1 percent (%) per year during the treatment period and for at least 6 months after the last dose of study drug
* Distant metastatic, recurrent or persistent squamous cell carcinoma, adenosquamous carcinoma or adenocarcinoma of the cervix that is not amenable to curative treatment with surgery and/or radiation therapy
* Either measurable or non-measurable disease. If disease is non-measurable or limited to the radiation field, a biopsy or fine-needle aspiration is required to confirm malignancy
* Eligible for carboplatin and paclitaxel chemotherapy in accordance with local standards of care
* Adequate hematological, renal and hepatic function
* Normal blood coagulation parameters
* Recovered (to Grade less than or equal to [<=] 1) from the effects of prior surgery, radiation therapy or chemoradiotherapy

Exclusion Criteria:

* Pregnant or lactating
* History of other malignancy within 5 years before screening, except for non-melanoma skin carcinoma
* Ongoing disease involving the bladder or rectum at screening/baseline. In participants with pelvic disease, absence of tumor in the bladder or rectal mucosa must be demonstrated by magnetic resonance imaging (MRI) (preferred method, or endoscopy/cystoscopy if MRI is not easily accessible) within 28 days before enrolment
* Evidence of abdominal free air
* Bilateral hydronephrosis
* Untreated central nervous system (CNS) metastases
* Prior chemotherapy for recurrent, persistent or metastatic cervical cancer. Prior adjuvant or neoadjuvant chemotherapy for Stage I-IVA disease (i.e. for non-metastatic disease) is permitted if completed greater than (>) 6 months before first study dose
* Prior chemoradiation within the 3 months preceding first study dose
* Prior radiotherapy delivered using cobalt
* Prior or current bevacizumab or other anti-angiogenic treatment
* Requirement for treatment with any medicinal product that contraindicates the use of any of the study drugs, may interfere with the planned treatment, affects participant compliance or puts the participant at high risk for treatment-related complications
* Treatment with another investigational agent within 28 days or 2 investigational agent half-lives before first study dose
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days before the first dose of bevacizumab or anticipation of the need for major surgery during the course of study treatment
* Minor surgical procedure within 2 days before the first dose of study drug
* Any prior history of fistula or GI perforation
* Known hypersensitivity to bevacizumab or any of its excipients, Chinese hamster ovary cell products or other recombinant human or humanized antibodies to any planned chemotherapy
* Active GI bleeding or ulcer
* Uncontrolled hypertension
* Clinically significant active cardiovascular disease
* National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0, Grade greater than or equal to (>=) 2 peripheral vascular disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with GI Perforation/Fistula Events by Grade According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0 | Baseline up to 24 months
Percentage of Participants with GI-Vaginal Fistula Events by Grade According to NCI-CTCAE Version 4.0 | Baseline up to 24 months
Percentage of Participants with GU Fistula Events by Grade According to NCI-CTCAE Version 4.0 | Baseline up to 24 months

SECONDARY OUTCOMES:
Time to First GI Perforation/Fistula | Baseline up to 24 months
Time to First GI-Vaginal Fistula | Baseline up to 24 months
Time to First GU Fistula | Baseline up to 24 months
Dose Intensity (Ratio of Actual Dose Administered Versus Intended Dose) for Bevacizumab During the Treatment Period | Baseline up to 24 months
Dose Intensity (Ratio of Actual Dose Administered Versus Intended Dose) for Carboplatin During the Treatment Period | Baseline up to 24 months
Dose Intensity (Ratio of Actual Dose Administered Versus Intended Dose) for Paclitaxel During the Treatment Period | Baseline up to 24 months
Duration of Treatment for Bevacizumab | Baseline up to 24 months
Duration of Treatment for Carboplatin | Baseline up to 24 months
Duration of Treatment for Paclitaxel | Baseline up to 24 months
Percentage of Participants with Adverse Events (AEs) | Baseline up to 24 months
Percentage of Participants with Serious Adverse Events (SAEs) | Baseline up to 24 months
Percentage of Participants with Adverse Events of Special Interest (AESIs) | Baseline up to 24 months
Percentage of Participants with AEs Leading to Treatment Interruption or Permanent discontinuation | Baseline up to 24 months
Percentage of Deaths Causally Related to Treatment | Baseline up to 24 months
Progression-Free Survival (PFS) According to Response Evaluation Criteria for Solid Tumors (RECIST) Version 1.1 | Baseline up to 24 months
Overall Survival (OS) | Baseline up to 24 months
Percentage of Participants with a Best Overall Response of Complete Response (CR) or Partial Response (PR) According to RECIST Version 1.1 | Baseline up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (43):
- Centro Oncologico Riojano Integral (CORI), La Rioja, Argentina
- Brazil (4):
  - Hospital das Clinicas - UFMG, Belo Horizonte, Minas Gerais
  - Oncologica Brasil S/S LTDA - EPP, Belém, Pará
  - Instituto Nacional de Cancer - INCa; Pesquisa Clinica, Rio de Janerio, Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Bulgaria (2):
  - Complex Oncological Center - Plovdiv, EOOD, Plovdiv
  - MHAT Nadezhda, Sofia
- Colombia (2):
  - Oncomedica S.A., Montería
  - Oncólogos de Occidente, Pereira
- Clinica CIMCA, San José, Costa Rica
- France (2):
  - Centre Francois Baclesse; Urologie Gynecologie, Caen
  - Institut Gustave Roussy; Oncologie Medicale, Villejuif
- Greece (2):
  - Alexandras General Hospital of Athens; Oncology Department, Athens
  - IASO, Athens
- Italy (4):
  - Istituto Tumori Napoli;Unità Operativa Oncologia Medica Uro-Ginecologica, Napoli, Campania
  - Universita' Cattolica Del Sacro Cuore; Reparto Ginecologia Oncologica, Rome, Lazio
  - Istituto Nazionale dei Tumori; Divisione Oncologia Chirurgica e Ginecologica, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Oncologia Medica, Milan, Lombardy
- Mexico (3):
  - Consultorio de Medicina Especializada, México, Mexico CITY (federal District)
  - Instituto Nacional de Cancerologia; Oncology, Distrito Federal
  - Centro Oncologico Estatal ISSEMYM, Toluca
- Panama (2):
  - Centro Oncológico de Panamá, Panama City
  - Centro Hemato Oncologico Panama, Panama City
- Poland (4):
  - Bialostockie Centrum Onkologi, Bialystok
  - Centrum Onkologii Instytut im. M.Sklodowskiej-Curie; Klinika Ginekologii Onkologicznej, Krakow
  - Wielkopolskie Centrum Onkologii im. M. Sklodowskiej-Curie, Poznan
  - Centrum Onkologii - Instytut M.Sklodowskiej-Curie; Klinika Ginekologii Onkologicznej, Warsaw
- IPO do Porto; Servico de Oncologia Medica, Porto, Portugal
- Romania (2):
  - Centrul de Oncologie Sfantul Nectarie, Craiova
  - Regional Institute of Oncology Iasi, Iași
- Russia (2):
  - Russian Oncology Research Center n.a. N.N. Blokhin Dpt of Clinical Pharmacology and Chemotherapy, Moscow
  - St. Petersburg Oncology & Gynecology; City Clinical Oncology Dispensary, Saint Petersburg
- Institute for Onc/Rad Serbia, Belgrade, Serbia
- South Africa (2):
  - Wits Clinical Research, Johannesberg
  - University of Pretoria; Department of Medical Oncology, Pretoria
- Spain (6):
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Hospital Duran i Reynals; Oncologia, Barcelona
  - Centro Oncologico MD Anderson International Espana, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia
  - Hospital Universitario la Fe; Servicio de Oncologia, Valencia
- Turkey (Türkiye) (2):
  - Ankara Baskent University Medicine Faculty; Gynaecology, Ankara
  - Istanbul Uni of Medicine Faculty; Oncology Dept, Istanbul

REFERENCES:
- [Derived] Redondo A, Colombo N, McCormack M, Dreosti L, Nogueira-Rodrigues A, Scambia G, Lorusso D, Joly F, Schenker M, Ruff P, Estevez-Diz M, Irahara N, Donica M, Gonzalez-Martin A. Primary results from CECILIA, a global single-arm phase II study evaluating bevacizumab, carboplatin and paclitaxel for advanced cervical cancer. Gynecol Oncol. 2020 Oct;159(1):142-149. doi: 10.1016/j.ygyno.2020.07.026. Epub 2020 Aug 4. PMID 32763109